CLINICAL TRIAL: NCT05237050
Title: Evaluation of Sound Therapy in a Population of Women With Fibromyalgia Aged Between 30 and 60 Years
Acronym: SONOMYAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-CHITS-010; 2021-A02461-40 (Other: Id-RCB)
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Chronic pain; Sound therapy; Tuning fork
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sound therapy associated with relaxation (Experimental)
  Interventions: Other: Sound therapy associated with relaxation
- Relaxation alone (Active Comparator)
  Interventions: Other: Relaxation alone

INTERVENTIONS:
Other: Sound therapy associated with relaxation — Each patient will attend a total of 3 sessions of about 15 minutes each, once by week.
  Sessions will start with relaxation. Then, sound therapy will be delivered using weighted medical tuning forks which resonate at a specific frequency. At the end of the session, the patient will be invited to take a short rest.
  Arms: Sound therapy associated with relaxation
Other: Relaxation alone — Each patient will attend a total of 3 sessions of about 15 minutes each, once by week.
  The procedure will be exactly the same than the other arm (relaxation, rest time), but the operator will not activate any tuning fork (so there will be no sound delivered during the session).
  Arms: Relaxation alone

SUMMARY:
This study focusing on sound therapy in patients with fibromyalgia is a single-centre, prospective, randomized study which evaluates the improvement or not of painful symptoms following relaxation sessions with sound therapy.

DETAILED DESCRIPTION:
Sound therapy consists in sound use as therapy and appears to mitigate or even relieve some symptoms.

The SonoMyal study intends to compare the effects of relaxation sessions with sound therapy delivered by tuning forks to a control group who will benefit from relaxation sessions without tuning fork activation, in a population of women with fibromyalgia.

The treatment consists in one session per week during 3 weeks, for a total of 3 sessions. Questionnaires to assess pain, anxiety and the ability to let go will be completed by patients before the beginning of the first session and at the end of the last session.

The main objective of the study is to assess with a Visual Analogue Scale of pain if 3 relaxation sessions with sound therapy delivered by tuning forks can improve pain perception in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30 and 60
* Fibromyalgia diagnosed according to the criteria of the combined Widespread Pain Index (WPI) and the Symptom Severity Scale (SSS) of the American College of Rheumatology ; and this whatever the previous analgesic medication and whatever the symptomatology
* Able to express her consent prior to participation in the study
* Affiliated to or beneficiary of a social security regimen

Exclusion Criteria:

* Total deafness in one or both ears (patients with age-related presbycusis can be included)
* Pregnant women
* Patient under judicial protection (guardianship, curatorship...) or safeguard of justice

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Pain intensity according to a Visual Analogic Scale (VAS) | Up to 4 weeks
  The minimum value of the scale, corresponding to no pain at all, is 0 and the maximum value is 10. Pain intensity will be assessed before and after each session and will be compared between the two groups.

SECONDARY OUTCOMES:
Impact on quality of life by Fibromyalgia Impact Questionnaire (FIQ) | Up to 4 weeks
  For this questionnaire, the score is between 0 and 100. A higher score indicates more impact of the condition on patient life.
Anxiety assessed by State Trait Anxiety Inventory questionnaire (STAI) | Up to 4 weeks
  For "State" STAI : the minimum value is 20 and the maximum value is 80. Higher scores mean a worse outcome, high level of anxiety.
  For "Trait" STAI : the minimum value is 21 and the maximum 77. Higher scores mean a worse outcome, high level of anxiety.
Qualitative assessment scale of the fluency of consciousness (EQFC) | Up to 4 weeks
  For "State" EQFC : the minimum value is 48 and the maximum value is 80. Higher scores mean a better outcome, high level of fluency.
  For "Trait" EQFC : the minimum value is 48 and the maximum value is 80. Higher scores mean a better outcome, high level of fluency.
Experiential phenomenological interviews | 4 weeks
  Only for the group of patients randomized in Arm 1 "Sound therapy associated with relaxation".
  Based on guided introspection and allow the description of background experiences of consciousness.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel DIAS ALVES, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- Gap Hospital, Gap, Hautes Alpes, France

IPD SHARING:
Plan to Share IPD: No